CLINICAL TRIAL: NCT03982641
Title: A Plan for Evaluating Costs and Outcomes of Colorectal Surgery in Emilia-Romagna (Emilia-Romagna Surgical Colorectal Cancer Audit-ESCA)
Brief Title: Emilia-Romagna Surgical Colorectal Cancer Audit- ESCA
Acronym: ESCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST153.07
Record Dates: First submitted 2019-05-28; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Financial Benefit; Colorectal Cancer; Surgery; Auditing Activity
Keywords: colorectal cancer surgery; auditing activity; economical analysis; surgical performance indicators
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Colon surgery: patients diagnosed with colon cancer, who undergone at least one surgical procedure at one of participating hospitals during the observational period
  Interventions: Procedure: all colorectal cancer surgical procedures
- Rectal surgery: patients diagnosed with rectal cancer, who undergone at least one surgical procedure at one of participating hospitals during the observational period
  Interventions: Procedure: all colorectal cancer surgical procedures

INTERVENTIONS:
Procedure: all colorectal cancer surgical procedures — colorectal cancer surgical procedures

SUMMARY:
Focus of this project is to evaluate the possible financial benefit resulting from an optimization of surgical outcomes throughout a collaborative and systematic auditing activity.The primary objective of this analysis is to assess the employed resources by National Health System related to surgical activities for primary colorectal cancer during a collaborative and systematic auditing activity in 8 Surgical Units of Emilia-Romagna

DETAILED DESCRIPTION:
Focus of this project is to evaluate the possible financial benefit resulting from an optimization of surgical outcomes throughout a collaborative and systematic auditing activity.

The primary objective of this analysis is to assess the employed resources by National Health System related to surgical activities for primary colorectal cancer during a collaborative and systematic auditing activity in 8 Surgical Units of Emilia-Romagna. A project team composed by experts in colorectal cancer care will be created with the task of identifying the needed resources to allocate to the project and the set of administrative, economic and performance indicators to be measured during the project. A friendly, time-preserving dataset that includes all the items to be collected to measure established indicators will be developed. An analysis on costs and performance indicators will be conducted on colorectal procedures performed between 1 January 2019 and 31 December 2019 within the participating centers. From the second year auditing activity will be implemented among institutions of Emilia-Romagna. Analysis results obtained from the first year of collecting data will be used as a starting feedback report to implement the auditing activity dedicated to colorectal cancer. During the whole second year monthly feedback reports will be drafted and used for monitoring costs and performances outcomes of colorectal surgery procedures between 1 January 2020 and 31 December 2020.

At the end of the second year a final analysis will be performed to compare resources employed for colorectal cancer surgery between the first and second year. Economical and performance data will be collected.

Focusing on costs, the main sources to be used are administrative databases. Full in-hospital costs will be collected for each patient for the time interval between the day of admission for surgery and the following post-operative 90-days. The Diagnosis Related Groups (DRG) standardized payments will be used to calculate inpatient costs.

Another source for cost and performance information is the clinical chart (paper or electronic) in all its parts. The investigators will focus primarily on set of data, that potentially could contribute to define the cost of care on basis of post-operative pathway. Key performance indicators common to both colon and rectal surgery or specific for one of the two surgical procedure will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of malignant colorectal cancer;
* Underwent colorectal cancer surgery;

Exclusion Criteria:

• multiple synchronous primary tumours;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients diagnosed with malignant colorectal cancer, who undergone at least one surgical procedure at one of participating hospitals during the observational period will be collected
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
health care resources utilization (HCRU) | 90 day post surgery
  To identify the resources delivered to surgical patients. Resource are retrieved from administrative database.
Cost relate to HCRU | 90 day post-surgery
  To identify the significant cost drivers for the surgical management of colorectal cancer patients and to verify the impact on economic resource consumption of the systematic auditing activities. Costs are retrieved from adminatrative database.

SECONDARY OUTCOMES:
% of patients with post-operative complications | 180 days post surgery
  To assess the frequency of post-operative complications, unplanned re-interventions and re-admission. This outcome is measured from data collected in Case Report Form (CRF)
Rate of mortality at 30 days | 30 days post surgery
  To assess mortality rates at 30 days. This outcome is measured from data collected in CRF and from administrative database.
Rate of mortality at 90 days | 90 days post surgery
  To assess mortality rates at 90 days. This outcome is measured from data collected in CRF and from administrative database.
Rate of mortality at 180 days | 180 days post surgery
  To assess mortality rates at 180 days. This outcome is measured from data collected in CRF and from administrative database.
% of patients discussed in Multidisciplinary team meeting | 180 days post surgery
  To assess the number of patient discussed within a multidisciplinary team meeting before colon rectal surgery. This outcome is measured from data collected in CRF.
% of patients who underwent minimally invasive resection | 180 day post surgery
  To assess the number of minimally invasive resections. This outcome is measured from data collected in CRF.
Conversion rate | 180 day post surgery
  to assess the rate of conversion surgery. This outcome is measured from data collected in CRF.
% of patients with adequacy of lymph node sampling | 180 days post surgery
  To assess adequate intraoperative lymph node sampling of colorectal surgery. This outcome will be measured from data collected in CRF.
Rate of anastomosis | 180 days post surgery
  To assess the rate of anastomosis after low anterior resection vs terminal colostomy. This outcome will be measured from relative data collected in CRF.
Rate of Miles procedure | 180 days post surgery
  to assess the rate of Miles procedures in rectal cancer patients. This outcome is measured from data collected in CRF.
Quality of Total Mesorectal Excision: rate of positive Circumferential Resection Margin in patients with rectal cancer. | 180 days post surgery
  To assess the rate of positive Circumferential Resection Margin in rectal cancer patient. This outcome will be measured from data collected in CRF.
Rate of loop ileostomy in patients with rectal cancer | 180 days post surgery
  To assess the rate of loop ileostomy after rectal cancer resection. This outcome is measured from data collected in CRF.
% of patients with rectal cancer who underwent preoperative chemo-radiation therapy | 180 days post surgery
  To assess the appropriateness of preoperative chemo-radiation therapy in rectal cancer patients. This outcome is measured from data collected in CRF.
Rate of preoperative chemo-radiation therapy in patients with rectal cancer | 180 days post surgery
  To assess the rate of preoperative chemo-radiation therapy in rectal cancer patients. This outcome is measured from data collected in CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Mattia Altini, physician, Principal Investigator — IRST
Locations (9):
- Italy (9):
  - Istituto Scientifico Romagnolo per lo studio e la cura dei tumori, Meldola, FC
  - AUO Chirurgia Generale e D'Urgenza Ospedale M.Bufalini, Cesena, Forli-Cesena
  - AUO CHIRURGIA GENERALE OSPEDALE G. B. Morgagni- Pierantoni, Forlì, Forli-Cesena
  - Auo Chirurgia Generale Ospedale Degli Infermi, Faenza, Ravenna
  - AUO Chirurgia Generale Ospedale Umberto I, Lugo, Ravenna
  - AUO Chirurgia Generale Ospedale Ceccarini, Riccione, Rimini
  - AOU Chirurgia Generale Ospedale G. Da Saliceto, Piacenza
  - AUO Chirurgia Generale ed Urgenza Ospedale S. Maria delle Croci, Ravenna
  - Auo Chirurgia Generale Ospedale Degli Infermi, Rimini

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Massa I, Ghignone F, Ugolini G, Ercolani G, Montroni I, Capelli P, Garulli G, Catena F, Lucchi A, Ansaloni L, Gentili N, Danesi V, Montella MT, Altini M; ESCA Collaborative Group. Emilia-Romagna Surgical Colorectal Cancer Audit (ESCA): a value-based healthcare retro-prospective study to measure and improve the quality of surgical care in colorectal cancer. Int J Colorectal Dis. 2022 Jul;37(7):1727-1738. doi: 10.1007/s00384-022-04203-w. Epub 2022 Jul 2. PMID 35779080